CLINICAL TRIAL: NCT02337218
Title: Electrical Stimulation for Improving Balance in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Larry Lavery, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 062012-035
Record Dates: First submitted 2014-11-07; First posted 2015-01-13 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-07

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SENSUS Pain Management System (Active Comparator): Electrical stimulation device worn on the leg delivering a dose of 50 volts.
  Interventions: Device: SENSUS Pain Management System
- SENSUS Pain Management System - Sham (Sham Comparator): Electrical stimulation device worn on the leg and programmed to deliver no stimulation.
  Interventions: Device: SENSUS Pain Management System

INTERVENTIONS:
Device: SENSUS Pain Management System — An electrical stimulation device worn on a band around the leg. This device was determined to be non-significant risk by the FDA.

SUMMARY:
This is a double-blind randomized clinical trial. Both patients and the podiatrist that will evaluate and monitor study patients will be blinded to electrical stimulation application. The manufacturer of the units will be asked to not inform which patient received which unit. Each unit will be coded with a unique identification number, and the manufacturer units revealed their status, placebo or electric stimulation, only at the end of data collection for the last patient. Subsequently, the investigators could match the status of the identification numbers with the corresponding units to start analyzing the data. Patients that receive an activated electrical stimulation unit will receive a standard dose of 50 volts as described above.

The investigator will enroll a cohort of 80 diabetes (type II) patients with peripheral neuropathy (see section 6 for sample size justification). The diagnosis of diabetes mellitus will be based on World Health Organization criteria.(World-Health-Organization 1999). The inclusion and exclusion criteria are described in table III. The clinical assessments are described in table IV. The investigator will discuss the study design, duration, and its risks with potential subjects asked to participate. The participant will be provided with a consent form to read at their leisure. The investigator will be available to answer questions or provide more explanation as requested by potential participants and their family.

DETAILED DESCRIPTION:
There will be a total of five study visits required for each patient. There will be one scheduled visit for baseline evaluation and four additional visits at 2 weeks, 4 weeks, 6 weeks during treatment and 8 weeks (2 weeks post stopping the treatment). The baseline visit will involve completion of a standardized intake form, which will include pertinent demographics such as age, height, weight, education level, occupation, and comorbidities of the study patient (see Table IV). Several clinical assessments will be performed at baseline as well as at each study visit to evaluate severity of neuropathy and skin perfusion as described in the table IV.

Clinical Assessments Baseline Medical History: This will include: duration and type of diabetes, type of diabetes medication (insulin, oral, combination therapy, diet), previous history of foot ulcers, previous history of falls, amputation (toe, foot), lower extremity bypass, lower extremity angioplasty, Coronary artery bypass surgery, cardiac angioplasty, arthritis, liver disease, osteoporosis, malignancy, and bone tumors. The Kaplan co-morbidity index will be used to record disease severity. The New York Heart Association criteria will be used to classify congestive heart failure, and the National Kidney Foundation Disease Outcomes Quality Initiative Clinical Practice Guidelines for chronic kidney disease to stage kidney disease. Research staff will document all prescription and over-the-counter medications. Research staff will measure height and weight to determine body mass index (BMI).

Baseline Social Factors: Marital status, years of education, type of work, tobacco history (pack years, current smoker, current use of chewing tobacco, previous smoker, no tobacco history), drug history (current, previous history, no drug history), education, occupation, and alcohol history will be assessed.

Screening Test for frailty assessment: Fried Frailty Criteria: Weight loss >10 pounds in preceding year; Grip strength; Low levels of physical activity; 15 foot walk time; Exhaustion[13] Screening for cognitive problem: MMSE score [15] Foot questionnaire and foot exam

Baseline & each 2- week follow-up (week 2, week 4, week 6, and week 8):

Peripheral Neuropathy: Research staff will evaluate Vibration Perception Threshold (VPT) Testing to evaluate large fiber neuropathy Semmes-Weinstein monofilaments, and the Modified Neuropathy Disability Score. (Armstrong and Lawrence 1998) will be done. Research staff will assess light touch and pressure sensation at nine sites on each foot using 4, 10, 26, and 60 Semmes-Weinstein gram monofilaments. (Diamond, Mueller et al. 1989) The Modified Neuropathy Disability Score is a scored clinical examination that includes Achilles deep tendon reflex, pressure, vibration sensation and temperature sensation in both feet.

Pain: Visual Analogue Scale Gait test: 8 sensors will be attached to the legs and lower back using comfortable straps and will be asked to walk 20 meters on a flat surface, two times. A third 20 meter walk will be performed with an additional distractive cognitive task (counting -1). The 4th test will be fast walking. Walking performance (e.g., speed, cadence, and stability) and spatio-temporal parameters of gait (e.g., velocity, stride time, gait inter-cycle variability, double support, and gait initiation) will be measured.

Balance test: The BalanSensTM kinematic sensor will be attached to the legs and lower back and will be used to measure the variation of subject's center of mass measured by the Romberg protocol including double stance, semi-tandem, and full-tandem tests. Patients will be asked to stand straight, feet together, hands crossed for 30 seconds, 20 seconds, and 15 seconds respectively for double stance test, semi-tendem, and full tandem tests with eyes open and closed.

Baseline and 6 weeks follow-up Activity Monitoring: Spontaneous daily physical activity will be monitored in home environment for 2 days using PAMSysTM Removal log: participants will be asked to note the time off, time on, and reason for removal if the PAMSysTM is removed during the 2 day collection period.

Quality of life questionnaire: SF12 Other assessment Fall log: participant will receive a log and agree to call the study overseer in the event of a fall during the 4 weeks study period.

Other patient information: if it was available patients record including medical history, neurological exam results, and physical examination may be gathered from patient record after authorization of the subject (see form T504a). In addition, subject photograph or video during experiment may be taken after subject's authorization.

ELIGIBILITY:
Inclusion Criteria:

* Men or women (non pregnant) 18 years old or above
* Diagnosed for Diabetes Mellitus (type 2)* and ADA criteria Diabetes
* Evidence of peripheral neuropathy on neurologic examination
* Identified by our clinical staff examination and based on the criteria explained in -ADA statement
* Agreed to participate in this study and comply with instruction

Exclusion Criteria:

* Amputation and active ulcers or infection
* Cognitive deficits
* MMSE score of 24 or lower
* Unable to stand for more than 5 minutes (including symptomatic orthostatic hypotension or pain)
* Any clinically significant orthopedic, muscular, or peripheral vascular disorders that affect balance
* Alcohol or substance abuse within 6 months or major psychiatric disorder

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Lavery, DPM, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

REFERENCES:
- [Background] Wrobel JS, Najafi B. Diabetic foot biomechanics and gait dysfunction. J Diabetes Sci Technol. 2010 Jul 1;4(4):833-45. doi: 10.1177/193229681000400411. PMID 20663446
- [Background] Thakral G, Kim PJ, LaFontaine J, Menzies R, Najafi B, Lavery LA. Electrical stimulation as an adjunctive treatment of painful and sensory diabetic neuropathy. J Diabetes Sci Technol. 2013 Sep 1;7(5):1202-9. doi: 10.1177/193229681300700510. PMID 24124947
- [Background] Najafi B, Crews RT, Wrobel JS. A novel plantar stimulation technology for improving protective sensation and postural control in patients with diabetic peripheral neuropathy: a double-blinded, randomized study. Gerontology. 2013;59(5):473-80. doi: 10.1159/000352072. Epub 2013 Jul 16. PMID 23860103
- [Background] Aminian K, Najafi B, Bula C, Leyvraz PF, Robert P. Spatio-temporal parameters of gait measured by an ambulatory system using miniature gyroscopes. J Biomech. 2002 May;35(5):689-99. doi: 10.1016/s0021-9290(02)00008-8. PMID 11955509
- [Background] Najafi B, Aminian K, Loew F, Blanc Y, Robert PA. Measurement of stand-sit and sit-stand transitions using a miniature gyroscope and its application in fall risk evaluation in the elderly. IEEE Trans Biomed Eng. 2002 Aug;49(8):843-51. doi: 10.1109/TBME.2002.800763. PMID 12148823
- [Result] Najafi B, Horn D, Marclay S, Crews RT, Wu S, Wrobel JS. Assessing postural control and postural control strategy in diabetes patients using innovative and wearable technology. J Diabetes Sci Technol. 2010 Jul 1;4(4):780-91. doi: 10.1177/193229681000400403. PMID 20663438

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SENSUS Pain Management System | SENSUS Pain Management System - Sham
Started | 17 | 11
Completed | 17 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SENSUS Pain Management System | SENSUS Pain Management System - Sham | Total
Number analyzed (Participants) | 17 | 11 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (11) | 64 (10) | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 12 | 9 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Qatar | 17 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Balance Test (BalanSense Device)
Description: Postural control changes will be measured using the BalanSense device in subjects assigned to use the active Electrical Stimulation (intervention group) and subjects assigned to non-functional stimulator (sham group). Balance will be assessed for both groups at baseline and at each follow-up visit, weeks 2, 4, 6 and 8. Static balance and postural compensatory strategy will be assessed using the body worn sensor technology. Measurements taken with eyes closed and eyes open.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: degrees^2
Arm/Group | SENSUS Pain Management System | SENSUS Pain Management System - Sham
Number analyzed (Participants) | 17 | 11
degrees^2
  Ankle sway - eyes open | 1.54 (0.71) | 1.72 (1.4)
  Hip sway - eyes open | 1.76 (0.93) | 1.94 (1.45)
  Ankle sway - eyes closed | 2.94 (1.94) | 2.79 (1.72)
  Hip sway - eyes closed | 3.23 (2.13) | 3.17 (0.97)

2. Primary Outcome: Peripheral Neuropathy Measured by Vibration Perception Threshold (VPT) Testing
Description: We will evaluate Vibration Perception Threshold (VPT) Testing to evaluate large fiber neuropathy in the feet.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: volts
Arm/Group | SENSUS Pain Management System | SENSUS Pain Management System - Sham
Number analyzed (Participants) | 17 | 11
volts | 41 (7) | 40 (10)

3. Primary Outcome: Gait Test (LegSys System)
Description: 8 sensors will be attached to the legs and lower back using comfortable straps and will be asked to walk 20 meters on a flat surface, two times. A third 20 meter walk will be performed with an additional distractive cognitive task (counting -1). The 4th test will be fast walking. Walking performance (e.g., speed, cadence, and stability) and spatio-temporal parameters of gait (e.g., velocity, stride time, gait inter-cycle variability, double support, and gait initiation) will be measured at weeks 2, 4, 6 and 8.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | SENSUS Pain Management System | SENSUS Pain Management System - Sham
Number analyzed (Participants) | 17 | 11
meters per second
  Stride velocity | 0.87 (0.22) | 0.82 (0.21)
  Stride time | 1.26 (0.14) | 1.35 (0.25)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | SENSUS Pain Management System | SENSUS Pain Management System - Sham
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/11
Other Adverse Events (participants affected / at risk) | 0/17 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT02337218/Prot_SAP_000.pdf